CLINICAL TRIAL: NCT06341777
Title: Telerehabilitation for Visual Field Defects: Clinical Efficacy of a Novel Multisensory Therapy for Adults and Children With Acquired Brain Lesions
Brief Title: Multisensory Telerehabilitation for Visual Field Defects
Acronym: MUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: IRCCS Fondazione Stella Maris (Other); Meyer Children's Hospital IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25M621
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Visual Field Defect Following Cerebrovascular Accident; Hemianopia; Brain Injuries
MeSH Terms: conditions — Hemianopsia; Brain Injuries | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Intervention (IM group) (Experimental): HVDFs patients who start the audio-visual telerehabilitation immediately
  Interventions: Behavioral: Audio-visual training (AVT) telerehabilitation
- WaitList Delayed Intervention (WL group) (Experimental): HVDFs patients waiting 1 month before receiving the audio-visual telerehabilitation.
  Interventions: Behavioral: Audio-visual training (AVT) telerehabilitation
- Healthy Participants (No Intervention): A group of 12 healthy participants is recruited for comparisons of MRI-based connectivity metrics

INTERVENTIONS:
Behavioral: Audio-visual training (AVT) telerehabilitation — Participants are trained at home, with remote supervision, for 3 weeks (5 days/week, 2 hours/day) using an audio-visual device suitable for telerehabilitation (AVDESK, Linari Medical). Specifically, visual stimuli (LEDs) appear on a semicircular panel, either alone or paired with an acoustic cues, at different eccentricities. Stimuli to the blind visual field (70%) and intact visual field (30%) are presented in random sequence. Patients are trained to scan the visual field by shifting their gaze (from the central fixation point) towards the visual target (with or without sounds), without head movements, and to report its presence by pressing the response key.
  Arms: Immediate Intervention (IM group); WaitList Delayed Intervention (WL group)

SUMMARY:
Brain injuries may cause the loss of the ability to see portions of the visual field, the so-called visual field defects (VFDs). VFDs significantly impact the survivors' functional recovery and quality of life, with the majority of patients displaying no spontaneous recovery or being left with residual deficits. Among the available therapies for VFDs, the compensatory scanning training is considered the most promising. Yet, current evidence is insufficient to recommend it in clinical practice, and the scientific community has stressed the need of more high-quality research. The present randomized clinical trial in patients with chronic VFDs caused by brain lesions aims at verifying the feasibility and efficacy of a novel telerehabilitation using a multisensory scanning therapy, by measuring its effects on visual functions and daily activities, and by looking for neural indicators of the therapy-induced improvements.

ELIGIBILITY:
Inclusion Criteria:

* Acquired homonymous visual field defect (HVFDs) due stroke, traumatic brain injury, tumor, surgery for epilepsy in a chronic stage of illness (time from the lesion >6 months)
* Normal hearing
* Normal or corrected-to-normal visual acuity

Exclusion Criteria:

* cognitive decline (adults)
* intellectual disability (children)
* major neurological or psychiatric disease
* being enrolled in another therapy for HVFDs

not being enrolled in another VFDs therapy.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Accuracy on the EF Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups]
  Computerized visual search task. Participants have to search for the target letter "F" surrounded by distractors "E"s. RTs: median search times (seconds) of correct responses.
Change from baseline in Response Times (RTs) on the EF Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups]
  Computerized visual search task. Participants have to search for the target letter "F" surrounded by distractors "E"s. RTs: median search times (seconds) of correct responses.
Change from baseline in Accuracy on the Triangle Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  Computerized visual search task. Participants have to report the number of triangles (targets) surrounded by square distractors. Accuracy: the proportion of correct responses (range 0-1)
Change from baseline in RTs on the Triangle Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  Computerized visual search task. Participants have to report the number of triangles (targets) surrounded by square distractors. RTs: median search times (seconds) of correct responses.
Change from baseline in RTs on the Numbers Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  Computerized visual search task. Participants have to point to numbers (1 to 15) in ascending order. RTs: median search times (seconds).
Change from baseline in omissions on the Bell Test (only children) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  Participants have to cross out Bells (targets) among different distractors. Omissions: number of omitted targets.
Change from baseline in RTs on the Bell Test (only children) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  Participants have to cross out Bells (targets) among different distractors. RTs: median search times (seconds).
Change from baseline in Accuracy on the Small Faces Test (only children) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  Participants have to cross out targets among distractors. Accuracy: the number of correct responses
Change from baseline in RTs on the Small Faces Test (only children) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  Participants have to cross out targets among distractors; RTs: median search times (seconds).

SECONDARY OUTCOMES:
Change from baseline in Daily Living Dependent on Vision Questionnaire (total score) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  A scale assessing the impact of HVFDs on nine activities of daily living. For each item, the score ranges from 0 ("No difficulty") to 4 ("Very frequent difficulties")
Change from baseline in the Reading test (reading time) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
Change from baseline in the Hamilton Anxiety Scale (total score; only adults) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  A scale assessing the presence of anxiety
Change from baseline in the Beck's Depression Inventory (BDI; total score; only adults) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  A scale assessing the presence of depressive symptoms
Change from baseline in the Multidimensional Anxiety Scale for Children (MASC; total score; only children) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  A scale assessing the presence of anxiety in children
Change from baseline in the Children Depression Inventory (CDI; total score; only children) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  A scale assessing the presence of depressive symptoms in children
Change from baseline in the visual field size (only adults) | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 6-month follow-ups
  Automated Humphrey Visual Field Analyzer.
Change from baseline in the amplitude of Visual Evoked Potentials (VEPs) | At baseline (at the beginning of the treatment), at the end of the treatment, and at the 6-month follow-up
Change from baseline in the latency of Visual Evoked Potentials (VEPs) | At baseline (at the beginning of the treatment), at the end of the treatment, and at the 6-month follow-up
Change from baseline in the connectivity of the Inferior Longitudinal Fasciculus | At baseline (at the beginning of the treatment) and at the end of the treatment
  High Angular Resolution Diffusion Imaging (HARDI) index of mean diffusivity
Change from baseline in the connectivity of the Superior Longitudinal Fasciculus | At baseline (at the beginning of the treatment) and at the end of the treatment
  High Angular Resolution Diffusion Imaging (HARDI) index of mean diffusivity
Change from baseline in the connectivity of the Inferior Fronto Occipital Fasciculus | At baseline (at the beginning of the treatment) and at the end of the treatment
  High Angular Resolution Diffusion Imaging (HARDI) index of mean diffusivity
Change from baseline in the connectivity of the Optic Radiations | At baseline (at the beginning of the treatment) and at the end of the treatment
  High Angular Resolution Diffusion Imaging (HARDI) index of mean diffusivity
Change from baseline in the connectivity of the Optic Tracts | At baseline (at the beginning of the treatment) and at the end of the treatment
  High Angular Resolution Diffusion Imaging (HARDI) index of mean diffusivity

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data will be made available on zenodo.com
Time Frame: Data will become available right before the first submission of the first paper.
Access Criteria: Upon request to l.diana@auxologico.it

REFERENCES:
- [Derived] Bolognini N, Diana L, Rossetti A, Melzi L, Basso G, Manzo V, Cruz-Sanabria F, Cammarata G, Cernigliaro F, Bianchi Marzoli S, Tinelli F, Fiori S, Casati C. Telerehabilitation for visual field defects with a multisensory training: a feasibility study. J Neuroeng Rehabil. 2025 Feb 24;22(1):34. doi: 10.1186/s12984-025-01573-4. PMID 39994637